CLINICAL TRIAL: NCT04620005
Title: Impact of Extra Corporal Membrane Oxygenation Services on Burnout Development in Intensive Care Units.
Acronym: burnout
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-20-113
Record Dates: First submitted 2020-10-20; First posted 2020-11-06 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2020-10

CONDITIONS: Burnout, Caregiver; Extracorporeal Membrane Oxygenation Complication; Intensive Care Unit
Keywords: burnout; Extracorporeal Membrane Oxygenation; Intensive care unit
MeSH Terms: conditions — Caregiver Burden; Burnout, Psychological | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO: The first group will include practitioners who work in intensive care unit with ECMO services
  Interventions: Other: Observational
- Non-ECMO: The second group will include practitioners who work in non-ECMO inventive care unit
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Survey

SUMMARY:
The burnout phenomenon first came to clinical science 50 years ago. It is exponentially rising worldwide which prompted its discoverers to develop the most popular tool for its assessment, known as the Maslach burnout inventory (MBI)1. Common symptoms of burnout include depression, irritability, and insomnia. The growing demand for extra-corporeal membrane oxygenation (ECMO) may have an effect on burnout as the newly introduced services is demanding in effort and put the practitioners on complex ethical and administrative situations.

We conducted a cross-sectional descriptive study using a combined methodological quantitative and qualitative approach involving a convenience sample of 1000 healthcare practitioners within surgical and medical ICUs of Hamad Medical Corporation (HMC), Qatar. We will use used two main instruments to develop an online questionnaire: - The MBI-human service survey (MBI-HSS) and the Leadership scale Expectations: we expect that we will have a new insight about the impact of these complex interventions on practitioner's burnout.

DETAILED DESCRIPTION:
This study predominates at investigating the BOS in ECMO ICU and non-ECMO ICU, and whether the leadership attitude could have effect on the mentioned syndrome problem.

Methodology Settings This study will in a tertiary hospital in the Middle East "Hamad Medical Corporation" as a main centre, the study will be disseminated an online survey among other centres who will agree to participate on. The participants will be screened for socio-demographic data such as age, gender, profession, marital state, education, native country, years of experience, weekly working hours and salary. The questionnaire was clarified to the potential respondents in order to clear any poor understanding. English used as the official language in the organization; translation of the used instruments to individual mother languages is not required.

Design Cross-sectional descriptive survey with purposeful sampling. Mixed qualitative and quantitative methodology used in this dissertation. Invitations to participate through the mail, anonymous questionnaire survey will be presented to the staff members including physicians, nurses and respiratory therapists who work as full time.

1. Study Population and Study Setting/ Location In this section describe the study population that is to be enrolled in the study, planned recruitment number and Inclusion and Exclusion Criteria to be listed here. Also list the Hospitals in which this study will be conducted ( e.g. HGH, Rumailah etc) The study population would include physicians, nurses, and respiratory therapists working in ICUs. The inclusion criteria will include practitioners working in intensive care unit including physician, respiratory therapists and nurses who agree to participate in the survey. We will exclude practitioners who decline to participate and who will not complete the questionnaires. A flow diagram will be prepared for the enrollment.

The participants will be approached through communication with one representative within the assigned ICUs within Qatar, in case of agreement we will ask for a list of mails from each department to be enrolled in the study.

1. Study procedures

The study will be conducted for 12 months from the time of ethical approval. Instrumentation

The used instrumentation is questionnaire that is divided into the following sections:

A) Condition of work effectiveness questionnaire (CWEQ): This scale consisted of 19 items developed by Kanter, (1977) measured by a 5-point Likert type response. (9) B) Maslach Burnout Inventory human services survey (MBI-HSS): The scale is a standardized instrument to measure burnout it utilize 9 items related to emotional exhaustion and it is most frequently used in health care researches, the nine items are calculated to get the whole score, scores of 27 and more signals severe burnout. (10) The percentage of high degree of burnout was used for advanced analysis. We will get permission to use this scale from (Mindgarden.com, USA) C) Leadership Behaviours scale (LS): The staff discernment of managers' leadership attitude will be measured using the 11 item Manager Action Scale. (11)

The questionnaires will be submitted in English form; no need for translation, as health care practitioners in the organization, must practice English that is the official language at workplace. The results of the analysis will be presented using descriptive methods. The quantitative and qualitative data will be analysed statistically, the relations between the variables will be interpreted, the relation between burnout score and socio-demographic variables, occupational stress score, and empowerment scale will be assessed statistically using (t-test, analysis of variance, correlation efficient and regression).

Ethical Considerations:

Participant identity kept confidential, final report would not contain any identity. Comprehensive explanation for the participants about the questionnaires, the type, purpose of the study and outcome was done, early rejection, or late withdrawal was permissive. Ethical approval was obtained according to the corporate regulations. The ethical consent attached after being approval from the medical research centre.

Health care practitioners working on ICU whether providing ECMO services or not will be eligible to participate in the study

The primary objective will be to detect the prevalence of burnout among health care practitioner s working in ICU with ECMO services The secondary objectives will be to compare the burnout association in ECMO and non ECMO ICU, the effect of leadership attitude on burnout syndrome and to look at the burnout in special population within the groups like respiratory therapists

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria will include practitioners working in intensive care unit including physician, respiratory therapists and nurses who agree to participate in the survey

Exclusion Criteria:

* practitioners who decline to participate and who will not complete the questionnaires.

  * Non ICU practitioners
  * Perfusionists

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - The study population would include physicians, nurses, and respiratory therapists working in ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire assessing prevalence of burnout among health care practitioners working in ICU with ECMO services | 1 year

SECONDARY OUTCOMES:
The difference in burnout association in practitioners in ICU with ECMO services and in conventional ICU | 1 year
effect of leadership attitude on burnout syndrome | 1 year
  Through specific questionnaire
burnout in special population within the respiratory therapists | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad medical corporation, Doha, DA, Qatar

IPD SHARING:
Plan to Share IPD: No
The identification and other details will be kept confidential as per our organization rules

REFERENCES:
- [Result] Moss M, Good VS, Gozal D, Kleinpell R, Sessler CN. An Official Critical Care Societies Collaborative Statement: Burnout Syndrome in Critical Care Health Care Professionals: A Call for Action. Am J Crit Care. 2016 Jul;25(4):368-76. doi: 10.4037/ajcc2016133. PMID 27369038
- [Result] Poncet MC, Toullic P, Papazian L, Kentish-Barnes N, Timsit JF, Pochard F, Chevret S, Schlemmer B, Azoulay E. Burnout syndrome in critical care nursing staff. Am J Respir Crit Care Med. 2007 Apr 1;175(7):698-704. doi: 10.1164/rccm.200606-806OC. Epub 2006 Nov 16. PMID 17110646
- [Result] Mealer M, Burnham EL, Goode CJ, Rothbaum B, Moss M. The prevalence and impact of post traumatic stress disorder and burnout syndrome in nurses. Depress Anxiety. 2009;26(12):1118-26. doi: 10.1002/da.20631. PMID 19918928
- [Result] Omar AS, Elmaraghi S, Mahmoud MS, Khalil MA, Singh R, Ostrowski PJ. Impact of leadership on ICU clinicians' burnout. Intensive Care Med. 2015 Nov;41(11):2016-7. doi: 10.1007/s00134-015-4008-6. Epub 2015 Aug 8. No abstract available. PMID 26254014
- [Result] Chuang CH, Tseng PC, Lin CY, Lin KH, Chen YY. Burnout in the intensive care unit professionals: A systematic review. Medicine (Baltimore). 2016 Dec;95(50):e5629. doi: 10.1097/MD.0000000000005629. PMID 27977605
- [Derived] Omar AS, Labib A, Hanoura SE, Rahal A, Kaddoura R, Chughtai TS, Karic E, Shaikh MS, Hamad WJ, ElHassan M, AlHashemi A, Khatib MY, AlKhulaifi A. Impact of Extracorporeal Membrane Oxygenation Service on Burnout Development in Eight Intensive Care Units. A National Cross-Sectional Study. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt B):2891-2899. doi: 10.1053/j.jvca.2022.02.018. Epub 2022 Feb 18. PMID 35300897
- [Derived] Omar AS, Hanoura S, Labib A, Kaddoura R, Rahhal A, Al-Zubi MM, Galvez RD, Shiju S, Al Jonidi MJ, Ragab H, Al Hashemi AA, Alumlla A. Burnout among Respiratory Therapists and Perception of Leadership: A Cross Sectional Survey Over Eight Intensive Care Units. J Intensive Care Med. 2022 Dec;37(12):1553-1562. doi: 10.1177/08850666221086208. Epub 2022 Mar 14. PMID 35285747